CLINICAL TRIAL: NCT07290595
Title: Comparative Analysis Of Dexmedetomidine And Dexamethasone As An Adjuvant To 0.5%Ropivacaine On Onset Of Ultrasound Guided Supraclavicular Brachial Plexus Block In Patients Undergoing Upper Limb Surgeries
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sahiwal medical college sahiwal (Other Government)
Responsible Party: Principal Investigator, Maryam Maqsood, Post-Graduate Resident, Sahiwal medical college sahiwal
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 173-IRB/SLMC/SWL
Record Dates: First submitted 2025-12-16; First posted 2025-12-18 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Post Operative Analgesia; Bradycardia; Hypotension; Upper Limb Surgeries
MeSH Terms: conditions — Bradycardia; Hypotension | interventions — Ropivacaine; Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Group A will receive 28ml of 0.5%Ropivacaine + 1mcg/kg Dexmedetomidine (diluted in 2ml normal saline) and Group B will receive 28ml of 0.5%Ropivacaine + 8mg Dexamethasone (2ml).
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group A (Other): 0.5%Ropivacaine + 1mcg/kg Dexmedetomidine
  Interventions: Drug: Ropivacaine + Dexmedetomidine
- Group B (Other): 0.5%Ropivacaine + 8mg Dexamethasone
  Interventions: Drug: Ropivacaine + dexamethasone

INTERVENTIONS:
Drug: Ropivacaine + Dexmedetomidine — Supraclavicular brachial plexus block will be performed under aseptic measures with the patient lying supine with head turned 30 degrees toward the contralateral side. A linear 7-13 MHz ultrasonography probe (ACUSON P500, digital color doppler ultrasound Siemens Germany) will be placed in supraclavicular fossa and slightly angled towards the thorax. The brachial plexus appears as multiple hypoechoic disks just superficial and lateral to the subclavian artery. After identification of brachial plexus, the proposed puncture site will be infiltrated with 1ml of 2% lignocaine. Then, 25-gauge spinal needle will be inserted using in plane technique, from lateral to medial direction until the tip is visualized near the brachial plexus. After careful aspiration for blood, 28ml of 0.5%Ropivacaine + 1mcg/kg Dexmedetomidine (diluted in 2ml normal saline) will be injected in 5ml increments to obtain uniform spread around brachial plexus
  Other Names: Supravlavicular Brachial Plexus Block with Ropivacaine and Dexmedetomidine
  Arms: Group A
Drug: Ropivacaine + dexamethasone — Supraclavicular brachial plexus block will be performed under aseptic measures with the patient lying supine with head turned 30 degrees toward the contralateral side. A linear 7-13 MHz ultrasonography probe (ACUSON P500, digital color doppler ultrasound Siemens Germany) will be placed in supraclavicular fossa and slightly angled towards the thorax. The brachial plexus appears as multiple hypoechoic disks just superficial and lateral to the subclavian artery. After identification of brachial plexus, the proposed puncture site will be infiltrated with 1ml of 2% lignocaine. Then, 25-gauge spinal needle will be inserted using in plane technique, from lateral to medial direction until the tip is visualized near the brachial plexus. After careful aspiration for blood,28ml of 0.5%Ropivacaine + 8mg Dexamethasone (2ml)will be injected in 5ml increments to obtain uniform spread around brachial plexus
  Other Names: Supraclavicular Brachial Plexus Block with Ropivacaine and Dexamethasone
  Arms: Group B

SUMMARY:
To compare the efficacy of dexmedetomidine and dexamethasone as an adjuvant to 0.5%ropivacaine on onset of ultrasound guided supraclavicular brachial plexus block in patients undergoing upper limb surgeries.

Ropivacaine hydrochloride, a long acting local anesthetic, is commonly used for supraclavicular block owing to its favorable safety profile especially in terms of minimal cardiotoxicity and less motor block. Dexmedetomidine, a highly selective alpha-2 adrenergic agonist, enhances the quality of supraclavicular block by providing sedation and analgesia while potentially prolonging the duration of block through hyperpolarization of nerve fibers. While, Dexamethasone, a synthetic corticosteroid with potent anti-inflammatory and immunosuppressive properties, prolongs duration of analgesia by reducing perineural inflammation and inhibiting nociceptive signal transmission. Supraclavicular brachial plexus block offers dense anesthesia for surgical procedures at or distal to the elbow with relatively high success rate, once described as "spinal of the arm". Moreover, supraclavicular brachial plexus block is an excellent alternative to general anesthesia in upper limb surgeries.

DETAILED DESCRIPTION:
After preparation, patients will be randomized into two groups of 33 each, where group A will receive 28ml of 0.5%Ropivacaine + 1mcg/kg Dexmedetomidine (diluted in 2ml normal saline) and group B will receive 28ml of 0.5%Ropivacaine + 8mg Dexamethasone (2ml). Anesthetist involved in drug administration and observation will be blinded to coded drugs prepared by another anesthetist who will not be involved further in the study. A detailed history will be taken regarding mode of injury, any pre-existing disease and previous surgery followed by local examination of patient will be done to rule out any systemic disease. On shifting to the operation theatre, standard monitoring like pulse-oximeter, electrocardiogram and non-invasive blood pressure measurement will be started. Supraclavicular brachial plexus block will be performed under aseptic measures with the patient lying supine with head turned 30o toward the contralateral side. A linear 7-13 MHz ultrasonography probe (ACUSON P500, digital color doppler ultrasound Siemens Germany) will be placed in supraclavicular fossa and slightly angled towards the thorax. The brachial plexus appears as multiple hypoechoic disks just superficial and lateral to the subclavian artery. After identification of brachial plexus, the proposed puncture site will be infiltrated with 1ml of 2% lignocaine. Then, 25-gauge spinal needle will be inserted using in plane technique, from lateral to medial direction until the tip is visualized near the brachial plexus. After careful aspiration for blood, study drugs will be injected in 5ml increments to obtain uniform spread around brachial plexus. Patient will be assessed every 5 minutes till complete sensory and motor block or for 30 minutes, whichever is earlier, using three point scale with pin prick technique for sensory block and modified bromage scale for motor block. Side effects and complications of the technique and drugs will be monitored and appropriately treated. Outcome of study will be to compare the time of onset of sensory and motor block between 2 groups.

ELIGIBILITY:
Inclusion Criteria

* Patients scheduled for upper limb surgery below mid-humerus level
* Patients aged 18 to 70 years
* Patients with ASA class I, II and III
* Male and non-pregnant females Exclusion Criteria
* Patients refusal
* Patients with pre-existing peripheral neuropathy of the upper limb
* Patients with the Infection at block site
* Patients with history of ischemic heart disease
* Patients with bleeding disorder or deranged coagulation profile
* Patients with known history of allergy to local anaesthetic or any other drugs used

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-01-13 (Actual); Primary Completion 2026-02-12 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Post Operative Analgesia | from performance of Block upto 5 minutes
  Onset of Sensory Block
Post Operative Analgesia | from performance of block upto 5 minutes
  Onset of Motor Block

CONTACTS AND LOCATIONS:
Overall Officials: Adeel Riaz, MD, Study Director — Sahiwal medical college sahiwal
Locations (1):
- Sahiwal Medical College, Sahiwal, Sāhīwāl, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Yes
Data will be available on request after completion of study i.e. March 2026
Supporting Information: Study Protocol, SAP, ICF
Time Frame: March 2026
Access Criteria: On Demand